CLINICAL TRIAL: NCT02364141
Title: Trunk Restraint Therapy: the Continuous Use of the Harness Could Promote Feedback Dependence in Post-stroke Patients. A Randomized Trial.
Brief Title: Trunk Restraint Therapy in Post-stroke Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Roberta de Oliveira Cacho, PhD, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 06/61199-5
Record Dates: First submitted 2015-02-05; First posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Stroke
Keywords: stroke; upper extremity; motor learning; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trunk restraint therapy (Experimental): Reaching training with trunk restraint by a harness that limited the trunk movements.
  Interventions: Other: Trunk restraint therapy
- Trunk unrestraint therapy (Active Comparator): Unrestraint reaching training, only with verbal feedback to maintain the trunk right position.
  Interventions: Other: Trunk unrestraint therapy

INTERVENTIONS:
Other: Trunk restraint therapy — Reaching training with trunk restraint by a harness that limited the trunk movements.
  Forty-five training minutes, twice a week, totaling twenty sessions, were performed. The training was based in the motor learning concepts including repetitive and task-specific practice. The training task consisted of grasping a cone (3.5 cm diameter base, 13 cm high) and fitting random targets as requested by the therapist in a training platform (54 cm length, 64 cm extent, 1.5 cm high) with 9 targets (6.5 cm diameter) placed 10-13 cm apart, along 3 lines. The targets that were ordered in a way that stimulated the complete range of motion of shoulder and elbow, had pictures, colors, letters and numbers on them yielding variability and feedback to the performing tasks.
  Arms: Trunk restraint therapy
Other: Trunk unrestraint therapy — Unrestraint reaching training, only with verbal feedback to maintain the trunk right position.
  Forty-five training minutes, twice a week, totaling twenty sessions, were performed. The training was based in the motor learning concepts including repetitive and task-specific practice. The training task consisted of grasping a cone (3.5 cm diameter base, 13 cm high) and fitting random targets as requested by the therapist in a training platform (54 cm length, 64 cm extent, 1.5 cm high) with 9 targets (6.5 cm diameter) placed 10-13 cm apart, along 3 lines. The targets that were ordered in a way that stimulated the complete range of motion of shoulder and elbow, had pictures, colors, letters and numbers on them yielding variability and feedback to the performing tasks
  Arms: Trunk unrestraint therapy

SUMMARY:
The aim of this study was to evaluate the long-term effects of the task-specific training with trunk restraint comparing to the free one in post-stroke reaching movements. Twenty hemiparetic chronic stroke patients were selected and randomized into two training groups: Trunk restraint group - TRG (reaching training with trunk restraint) and Trunk free group - TFG (unrestraint reaching). Twenty sessions with forty-five minutes of training were accomplished. The subjects were evaluated in pre-treatment (PRE), post-treatment (POST) and three months after the completed training (RET). The measures administered were the Modified Ashworth Scale, Barthel Index, Fugl-Meyer Scale and kinematic analysis (movement trajectory, velocity, angles).

DETAILED DESCRIPTION:
Twenty stroke subjects were recruited from the Physiotherapy and Occupational Therapy Outpatient Unit of the University Hospital at Campinas - UNICAMP and all of them signed informed consent forms previously approved by the Research Ethics Committee of the University (#110/2004). Ten healthy subjects were also selected to obtain normal reference parameters of kinematic assessment. Patients had sustained a single and chronic (>6 months post-event) unilateral stroke of non-traumatic origin, with hemiparetic sequel in the upper limb, could understand simple instructions, perform community gait, and had a good sitting balance. Those with shoulder pain or other neurological and orthopedic conditions affecting the reaching movement ability or trunk, hemispatial neglect or apraxia were excluded. The patients who met the inclusion criteria were stratified to one of two groups. A sealed opaque envelope containing a single cheat of paper marked with numbers 1 (group 1) or 2 (group 2), was used to allocate the patient. This procedure was made by an external assessor. The patients were not informed about the different treatment groups and therefore, they were blind for the type of intervention applied.

The muscle tone (shoulder and elbow flexors) was evaluated using the Modified Ashworth Scale (MAS)9; motor impairment was evaluated using the upper limb section of Fugl-Meyer Assessment Scale (FM) and activities of daily living was assessed by the Barthel Index (BI). Kinematic data were recorded by an infrared system of motion analysis (Qualisys Motion Capture System - 2.57 Sweden) with sample frequency of 240 Hz, during 8 seconds. The coordinated data was low-pass filtered using a 6 Hz, finite impulse response filter with order 26 using the Matlab software. Five infrared reflexive markers were used. For the kinematic capture, the subjects were seated in a chair and invited to fit a cone in a target placed within arm's length (measured on the non-affected arm from the medial border of axilla to the distal wrist crease). The target was placed so that only the arm movement was required to reach the target. The initial hand position of the affected arm was on the lateral trunk, with the shoulder in neutral position and the elbow close to the side of the body (90°). Three trials of 6 to 8 seconds' time were recorded and a media was used to calculate the evaluated data.From the collected dates, values concerning to sagittal (YZ), horizontal (XY) and 3-dimensional (XYZ) planes were computed.

Trunk displacement was verified in millimeters as sagittal movement of marker 3.

Index of curvature was measured from marker 5. This index shows the straightness of the wrist trajectory from the initial position to the goal, resulting in a ratio of actual end point path to a straight line (index = 1, whereas a semicircle has an index of 1.57).

Shoulder angles were calculated using 2 vectors formed from marker 1 to marker 2, and from marker 2 to marker 4; with flexion/extension movements in sagittal plane and adduction/abduction movement in horizontal plane. Full horizontal abduction and the anatomical position were considered at 0°. Flexion/extension elbow angles were measured using 2 vectors formed from marker 2 to 4 and from marker 4 to 5, using the sagittal and horizontal planes. The elbow full extension was considered at 180°.

Movement time was defined as differences between movement onsets and offsets which tangential velocity rose above and fell below at 5% of its peak value.

The maximum tangential velocity of the arm was computed from the velocity vector expressed by a numerical differentiation from wrist and sternum markers in the 3-dimensional plane. Numbers of peaks and the percentage of movement time at the maximum peak velocity (rate - %) were extracted from tangential velocity traces.

The evaluations were performed by a blind researcher, in admission time (PRE), after the end of the twenty treatment sessions (POST) and three months after the training was completed (retention test - RET).

The selected patients were randomized individually into two training groups:

Trunk restraint group - TRG (n = 10): reaching training with trunk restraint by a harness that limited the trunk movements.

Trunk free group - TFG (n = 10): unrestraint reaching training, only with verbal feedback to maintain the trunk right position.

Forty-five training minutes, twice a week, totaling twenty sessions, were performed (The participants will be trained for 10 weeks, and with 3 months of follow-up).

The training was based in the motor learning concepts including repetitive and task-specific practice. The training task consisted of grasping a cone (3.5 cm diameter base, 13 cm high) and fitting random targets as requested by the therapist in a training platform (54 cm length, 64 cm extent, 1.5 cm high) with 9 targets (6.5 cm diameter) placed 10-13 cm apart, along 3 lines. The targets that were ordered in a way that stimulated the complete range of motion of shoulder and elbow, had pictures, colors, letters and numbers on them yielding variability and feedback to the performing tasks.

Chi-squared, or Fisher's tests, was used to compare the categorical variables (i.e. gender) between the three groups (HS, TRG, TFG). Mann-Whitney (for two groups) and Kruskal-Wallis (for three groups) tests were used to compare the ratio dates (i.e. age, years since stroke) measured at a single instant. Repeated-measure analysis of variance (ANOVA) and appropriate post-hoc tests (Bonferroni) were applied to compare the numerical variables (i.e. kinematics dates) between groups and instants. The normality of the kinematic variables was detected by Shapiro-Francia test and for variables that were not normal was proposed Box-Cox transformation. The significance level adopted for the statistical tests was 5% (p< 0.05).

ELIGIBILITY:
Inclusion Criteria:

* single and chronic (>6 months post-event) unilateral stroke of non-traumatic origin
* hemiparetic sequel in the upper limb
* could understand simple instructions
* perform community gait
* had a good sitting balance

Exclusion Criteria:

* shoulder pain or other neurological and orthopedic conditions affecting the reaching movement ability or trunk
* hemispatial neglect
* apraxia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-08; Primary Completion 2007-11 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
muscle tone (shoulder and elbow flexors) | 10 weeks
  by Modified Ashworth Scale (MAS)
upper limb motor impairment | 10 weeks
  by Fugl-Meyer Assessment Scale (FM)
activities of daily living level | 10 weeks
  by Barthel Index (BI)

SECONDARY OUTCOMES:
Trunk displacement in millimeters as sagittal movement | 10 weeks
  Kinematic data
Index of curvature of wrist trajectory | 10 weeks
  Kinematic data
Shoulder and elbow angles | 10 weeks
  Kinematic data
Movement time | 10 weeks
  Kinematic data
maximum tangential velocity | 10 weeks
  Kinematic data
Numbers of peaks | 10 weeks
  Kinematic data
maximum peak velocity | 10 weeks
  Kinematic data

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Borges, PhD, Study Director — University of Campinas, Brazil

REFERENCES:
- [Background] Cirstea MC, Levin MF. Compensatory strategies for reaching in stroke. Brain. 2000 May;123 ( Pt 5):940-53. doi: 10.1093/brain/123.5.940. PMID 10775539
- [Background] Archambault P, Pigeon P, Feldman AG, Levin MF. Recruitment and sequencing of different degrees of freedom during pointing movements involving the trunk in healthy and hemiparetic subjects. Exp Brain Res. 1999 May;126(1):55-67. doi: 10.1007/s002210050716. PMID 10333007
- [Background] Michaelsen SM, Levin MF. Short-term effects of practice with trunk restraint on reaching movements in patients with chronic stroke: a controlled trial. Stroke. 2004 Aug;35(8):1914-9. doi: 10.1161/01.STR.0000132569.33572.75. Epub 2004 Jun 10. PMID 15192250
- [Background] Michaelsen SM, Luta A, Roby-Brami A, Levin MF. Effect of trunk restraint on the recovery of reaching movements in hemiparetic patients. Stroke. 2001 Aug;32(8):1875-83. doi: 10.1161/01.str.32.8.1875. PMID 11486120
- [Background] Michaelsen SM, Dannenbaum R, Levin MF. Task-specific training with trunk restraint on arm recovery in stroke: randomized control trial. Stroke. 2006 Jan;37(1):186-92. doi: 10.1161/01.STR.0000196940.20446.c9. Epub 2005 Dec 8. PMID 16339469
- [Background] Woodbury ML, Howland DR, McGuirk TE, Davis SB, Senesac CR, Kautz S, Richards LG. Effects of trunk restraint combined with intensive task practice on poststroke upper extremity reach and function: a pilot study. Neurorehabil Neural Repair. 2009 Jan;23(1):78-91. doi: 10.1177/1545968308318836. Epub 2008 Sep 23. PMID 18812433
- [Background] Wu CY, Chen YA, Chen HC, Lin KC, Yeh IL. Pilot trial of distributed constraint-induced therapy with trunk restraint to improve poststroke reach to grasp and trunk kinematics. Neurorehabil Neural Repair. 2012 Mar-Apr;26(3):247-55. doi: 10.1177/1545968311415862. Epub 2011 Sep 8. PMID 21903975
- [Background] Stewart JC, Gordon J, Winstein CJ. Control of reach extent with the paretic and nonparetic arms after unilateral sensorimotor stroke: kinematic differences based on side of brain damage. Exp Brain Res. 2014 Jul;232(7):2407-19. doi: 10.1007/s00221-014-3938-5. Epub 2014 Apr 10. PMID 24718494
- [Result] de Oliveira R, Cacho EW, Borges G. Improvements in the upper limb of hemiparetic patients after reaching movements training. Int J Rehabil Res. 2007 Mar;30(1):67-70. doi: 10.1097/MRR.0b013e3280143bbf. PMID 17293723
- [Derived] de Oliveira Cacho R, Cacho EWA, Ortolan RL, Cliquet A Jr, Borges G. Trunk restraint therapy: the continuous use of the harness could promote feedback dependence in poststroke patients: a randomized trial. Medicine (Baltimore). 2015 Mar;94(12):e641. doi: 10.1097/MD.0000000000000641. PMID 25816031